CLINICAL TRIAL: NCT06872242
Title: Italian PheNotypes Obstructive Sleep Apnea Study
Acronym: IPNOS
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 09M205
Record Dates: First submitted 2025-02-28; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Sleep Apnea
Keywords: Sleep apnea; Phenotypes; Diagnosis
MeSH Terms: conditions — Sleep Apnea Syndromes; Disease | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspected obstructive sleep apnea (OSA): Patients referred to the Italian Sleep Centres because of suspected OSA
  Interventions: Diagnostic Test: Polysomnography

INTERVENTIONS:
Diagnostic Test: Polysomnography — Polysomnography after enrollment for suspected obstructive sleep apnea

SUMMARY:
Obstructive Sleep Apnea (OSA) is the most common sleep-related breathing disorder, representing a major socioeconomic burden on healthcare systems worldwide. Studies performed in Europe in the last twenty years showed a very high prevalence and highlighted that the severity of untreated OSA worsens over time. OSA is associated also with an increased risk to develop cardiovascular, cerebrovascular and metabolic diseases. Finally, recent studies reported a very high mortality in untreated OSA patients, including those with mild severity.

Data on European population have been obtained by the "ESADA group" (European Sleep Apnea Database) , a consortium of 25 sleep center across Europe that includes three Italian Research Hospitals. The ESADA showed significant differences between European geographical macrozones in terms of symptoms and complications. However, no data are available for the Italian population in terms of prevalence, clinical presentation and comorbidities.

The present project aims to overcome this limitation by obtaining a more defined picture of OSA in Italy. A cohort study was designed in collaboration with the Sleep Centers endorsed by the Italian Scientific Society of Sleep Medicine (AIMS).

Aims of the present project are to:

1. Assess the distribution different physiological (endotypes) and clinical patterns (phenotypes) of OSA in Italian patients
2. Analyze the association between OSA and co-morbidities
3. implementation of an "Italian database" for long-term follow-up studies.

Methods

* Clinical, sleep study and treatment data will be collected for each patient. A clinical questionnaire will be developed in order to standardize the clinical data collection; to this end a feasibility study will be performed on 100 patients (25 pts for Coordinator/HUB center).
* Excessive daytime Sleepiness, Neurocognitive, anxiety/depression screening
* A web-based data collection platform will be designed to store pseudo-anonymized individual data.

OUTCOMES

1. Distribution of OSA severity in Italy according to the different classification methods
2. Definition of metabolic, cerebro- and cardiovascular risk factors prevalence associated with OSA in Italian Population
3. Distribution of different physiological and clinical patterns and their association with co-morbidities
4. Definition of a screening/case finding questionnaire for Italian Population
5. Definition of an ongoing cohort of patients that will be followed-up
6. Implementation of an OSA registry that will be shared with Italian Health System or Agencies to designed preventive or early diagnosis interventions to reduce the health impact of the disease.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) is the most common sleep-related breathing disorder, representing a major socioeconomic burden on healthcare systems worldwide. Studies performed in Europe in the last twenty years showed a very high prevalence and highlighted that the severity of untreated OSA worsens over time. OSA is associated also with an increased risk to develop cardiovascular, cerebrovascular and metabolic diseases. Finally, recent studies reported a very high mortality in untreated OSA patients, including those with mild severity.

Data on European population have been obtained by the "ESADA group" (European Sleep Apnea Database), a consortium of 25 sleep center across Europe that includes three Italian Research Hospitals. The ESADA showed significant differences between European geographical macrozones in terms of symptoms and complications. However, no data are available for the Italian population in terms of prevalence, clinical presentation and comorbidities.

The present project aims to overcome this limitation by obtaining a more defined picture of OSA in Italy. A cohort study was designed in collaboration with the Sleep Centers endorsed by the Italian Scientific Society of Sleep Medicine (AIMS).

Aims of the present project are to:

1. Assess the distribution different physiological (endotypes) and clinical patterns (phenotypes) of OSA in Italian patients
2. Analyze the association between OSA and co-morbidities by taking into account the phenotypes already described in the literature, i.e., ESADA, Icelandic Sleep Cohort, and BAVENO classification;
3. implementation of an "Italian database" for long-term follow-up studies. The project will set an HUB and SPOKE organization that include 4 leading research Sleep Center distributed over the Italian territory in collaboration with the Italian Scientific Society of Sleep Medicine (AIMS) network. AIMS is member of the European Federation of National Sleep Society as well as part of World Sleep Association.

Methods

* Clinical, sleep study and treatment data will be collected for each patient. A clinical questionnaire will be developed in order to standardize the clinical data collection; to this end a feasibility study will be performed on 100 patients (25 pts for Coordinator/HUB center). Additional clinical tests will include: EKG, Spirometry, ABPM, standard blood chemistry, CPR, TSH reflex, glycemic control assesment, Vitamin D and B12.
* Excessive daytime Sleepiness, Neurocognitive, anxiety/depression screening will be performed by means of ESS, MOCA and HADS, respectively
* A web-based data collection platform will be designed to store pseudo-anonymized individual data.

OUTCOMES

1. Distribution of OSA severity in Italy according to the different classification methods (AHI based; hypoxic burden; Icelandic Sleep Cohort, ESADA and BAVENO method)
2. Definition of metabolic, cerebro- and cardiovascular risk factors prevalence associated with OSA in Italian Population
3. Distribution of different physiological and clinical patterns and their association with co-morbidities; analysis of differences with other populations.
4. Definition of a screening/case finding questionnaire for Italian Population
5. Definition of an ongoing cohort of patients that will be followed-up
6. Implementation of an OSA registry that will be shared with Italian Health System or Agencies to designed preventive or early diagnosis interventions to reduce the health impact of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Suspected Obstructive Sleep Apnea
* Age 18 years or older

Exclusion Criteria:

* Unstable psychiatric disease
* Limited life expectancy due to illness unrelated to sleep apnoea or other medical conditions which may interfere with the study protocol in the opinion of the investigator

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients referred to the Italian Sleep Centres because of suspected Obstructive Sleep Apnea
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-10-23 (Estimated); Study Completion 2025-10-23 (Estimated)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index | At enrollment
  Apnea-Hypopnea Index as determined by Polysomnography
Oxygen saturation | At enrollment
  Oxygen saturation as determined by Polysomnography

CONTACTS AND LOCATIONS:
Locations (30):
- Italy (30):
  - ASP Cosenza- PO Beato Angelico, Acri
  - AOU delle Marche, Ancona
  - AOU Policlinico di Bari, Bari
  - ASST Papa Giovanni XXIII, Bergamo
  - Casa di cura San Francesco-Istituto Madre Rubatto, Bergamo
  - AUSL Bologna - Clinica odontoiatrica DIBINEM, Bologna
  - AUSL Bologna - Ospedale di Bellaria, Bologna
  - AOU Cagliari - Centro interdipartimentale dei disturbi del sonno, Cagliari
  - AOU Rodolico-S. Marco, Catania
  - ASP Cosenza- P.O. di Rossano, Corigliano-Rossano
  - Distretto Sanitario Cosenza- Savuto- Ambulatorio di Medicina del Sonno, Cosenza
  - AOU Ospedali Riuniti di Foggia, Foggia
  - Opera Don Uva Universo Salute, Foggia
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Ospedale Carlo Urbani, Iesi
  - IRCCS Istituto Neurologico "Carlo Besta", Milan
  - Istituto Auxologico Italiano, Milan
  - Ospedale San Paolo, Milan
  - AO dei Colli - PO Monaldi, Napoli
  - Ospedali Riuniti Villa Sofia Cervello, Palermo
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - IRCCS Fondazione Mondino, Pavia
  - Istituti Clinici Scientifici Maugeri, Pavia
  - Casa di Cura "Villa Serena", Pescara
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - IRCCS Neuromed - Istituto Neurologico Mediterraneo, Pozzilli
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Policlinico Tor Vergata, Roma
  - AOU Città della Salute e della Scienza di Torino - SC Otorinolaringoiatria, Torino
  - USL Umbria1 - Ambulatorio disturbi del sonno, Umbertide

IPD SHARING:
Plan to Share IPD: No